CLINICAL TRIAL: NCT06736548
Title: Sleep Treatment Education Program Together (STEP-Together): An Online Group Educational Intervention for Insomnia in Cancer Survivors
Brief Title: Sleep Treatment Education Program for Cancer Survivors: STEP-Together
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christopher Recklitis, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-505
Record Dates: First submitted 2024-12-12; First posted 2024-12-16 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Insomnia; Insomnia Chronic; Survivorship
Keywords: Insomnia; Chronic Insomnia; Cancer Survivorship
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STEP-Together Intervention (Experimental): Enrolled participants will complete the educational intervention session (STEP-Together) delivered by an interventionist during an online group videoconference session.
  -Up to 12 participants will also take part in a coaching session 1 week after the virtual intervention session.
  Interventions: Behavioral: The Sleep Treatment Education Program Together (STEP-Together); Behavioral: Coaching Session

INTERVENTIONS:
Behavioral: The Sleep Treatment Education Program Together (STEP-Together) — STEP-Together is delivered in a single videoconference group session delivered live by a presenter. During the session, the participants are able to see and hear the presenter, view the presentation slides, and ask questions. The presentation includes educational information on the problem of insomnia after cancer and specific suggestions for improving sleep. Suggestions are presented in four sections addressing lifestyle issues, sleep environment, sleep timing, and managing expectations and challenges. During the course of the session, participants are asked to use these suggestions to develop an individual sleep action plan they will use to improve their sleep.
  Other Names: STEP-Together
Behavioral: Coaching Session — Coaching sessions are brief (<1hour) sessions intended to support participants in implementing their personal sleep self-management plan. In the session, participants are asked to review their progress with their plan, report on areas of sucess and difficulty with adoption, and to problem solve with the study team as needed to support their sucessful implementation their plan.

SUMMARY:
This single-arm research study of off-treatment cancer survivors with self-reported symptoms of insomnia will test the Sleep Treatment Education Program Together (STEP-Together) intervention which is delivered as a synchronous group session by videoconference.

DETAILED DESCRIPTION:
This single-arm research study of off-treatment cancer survivors with self-reported symptoms of insomnia will test the Sleep Treatment Education Program Together (STEP-Together) intervention which is delivered as a virtual group session.

The research study procedures including screening for eligibility and questionnaires.

Participation in this research study is expected to last about 16 weeks.

It is expected about 90 people will participate in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* History of a cancer diagnosis (except non-melanoma skin cancer) ≥ 6 months prior
* No active cancer therapy (excluding chemoprevention) in the past four months, and no further therapy planned.
* Significant insomnia as evidenced by an Insomnia Severity Index score ≥ 8
* Regular access to the internet
* Able to read and write in English

Exclusion Criteria:

* Usual bedtime does not fall between 5:00 pm and 5:00 am.
* Employment in a position where falling asleep at work could impact public safety (such as air traffic-controller, operating heavy machinery).
* Ever diagnosed with Bipolar Disorder or with Seizure Disorder, currently taking medications to prevent a seizure, or have experienced a seizure in the prior 12 months.
* Any impairment (e.g., hearing, visual, cognitive) that interferes with the ability to complete all study procedures independently.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) Score from Baseline to 8 weeks Post-Intervention | Baseline to 8 weeks post-intervention
  Assessed by the Insomnia Severity Index, a 7-item measure measuring insomnia over the previous two weeks with answers graded on a 5-point Likert scale, ranging from 0 "No Problem" to "4 "Very Severe" for a total score range of 0 to 28. A higher score reflects moderate to severe insomnia symptoms.

SECONDARY OUTCOMES:
Change in Total Mood Disturbance (TMD) Scale from the Profile of Mood States - Short Form (POMS-SF) Score from Baseline to 8 weeks Post-Intervention | Baseline to 8 weeks post-intervention
  Assessed by the POM-SF, a 35-item measure of feelings and mood over the 2 weeks prior to questionnaire administration. Answers are graded on a 5-point Likert scale, ranging from 0 "Not At All" to 4 "Extremely." A higher score reflects more negative moods and lower vigor.
Change in Perceived Cognitive impairment Scale from Baseline to 8 weeks Post-Intervention | Baseline to 8 weeks post-intervention
  Assessed by the Perceived Cognitive Impairment Scale, a 20-item measure with answers graded on a 5-point Likert scale, ranging from 0 "Never" to 4 "Several Times a Day" for a total score range of 0 to 80. A higher score indicates poorer functioning. This scale is found in the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-COG).
Change in Impact of Cognitive Function on Quality of Life Scale from Baseline to 8 weeks Post-Intervention | Baseline to 8 weeks post-intervention
  Assessed by the Impact of Cognitive Function on Quality of Life Scale, a 4-item measure with answers graded on a 5-point Likert scale, ranging from 0 "Not At All" to 4 "Very Much" for a total score range of 0 to 16. A higher score indicates better cognitive function and a lower impact on quality of life. This scale is found in the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-COG).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Recklitis, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu